CLINICAL TRIAL: NCT07066631
Title: The Pregnancy and Postpartum Mental Health Optimization Virtual Intervention Network (MOVIN): Randomized Controlled Trial
Brief Title: The Pregnancy and Postpartum Mental Health Optimization Virtual Intervention Network
Acronym: MOVIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other); The Ottawa Hospital (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CTO Project ID: 5038
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Depression; Postpartum; Anxiety; Pregnancy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Other): Access to online resources and educational materials about general mental health, maternal mental health, depression and anxiety in the pregnancy and postpartum period, and an up-to-date listing of treatment services available in Ontario. These resources are maintained by the MOVIN study team.
  Interventions: Other: Enhanced Usual Care
- MOVIN (Experimental): Enhanced Usual Care plus MOVIN Care Platform. The MOVIN Care Platform is virtual collaborative care intervention with a stepped care approach in which a care coordinator directs participants to one or more evidence-based virtual interventions as appropriate.
  Interventions: Other: MOVIN Care Platform; Other: Enhanced Usual Care

INTERVENTIONS:
Other: Enhanced Usual Care — Access to online resources and educational materials about general mental health, maternal mental health, depression and anxiety in the pregnancy and postpartum period, and an up-to-date listing of treatment services available in Ontario. These resources are maintained by the MOVIN study team.
  Arms: Enhanced Usual Care
Other: MOVIN Care Platform — Virtual collaborative care intervention with a stepped care approach in which a care coordinator directs participants to one or more evidence-based virtual interventions as appropriate.
  Arms: MOVIN
Other: Enhanced Usual Care — Access to online resources and educational materials about general mental health, maternal mental health, depression and anxiety in the pregnancy and postpartum period, and an up-to-date listing of treatment services available in Ontario. These resources are maintained by the MOVIN study team.
  Arms: MOVIN

SUMMARY:
Depression, anxiety, and related disorders such as post-traumatic stress and obsessive compulsive disorder affect about 20% of pregnant and postpartum people. When not treated properly, these issues negatively impact not only affected people, but also their children's health and development. Only 1 in 5 receive adequate treatment, so identifying new system-wide approaches to reliably deliver recommended care to perinatal mental health patients all is a crucial health care priority. The Pregnancy and Postpartum Mental health Optimization Virtual Intervention Network (MOVIN) is a scalable perinatal mental health platform building on the evidence-based Collaborative care delivery model. MOVIN's online platform allows patients to connect with a care coordinator to co-develop personalized treatment recommendations, in collaboration with their primary care clinician and a perinatal psychiatrist when needed; progress is tracked to re-evaluate.

DETAILED DESCRIPTION:
The Pregnant and Postpartum Mental Health Optimization Virtual Intervention Network (MOVIN) is a model of stepped, collaborative care delivered virtually, accessible to pregnant and postpartum individuals across Ontario based at Women's College Hospital. Access to MOVIN includes access to a web platform with curated educational material and treatment resources, personalized treatment planning between a participant and the MOVIN Care Coordinator (informed by systematic measurement-based follow-up of mental health symptoms), liaison between the MOVIN Care Coordinator and the participant's primary care clinician, and direct referral to a perinatal psychiatrist if required. Participants will be allocated 1:1 (intervention: control) using a computer-generated random allocation sequence in randomly varying block sizes. The primary outcome will be depressive symptoms (considered as a continuous variable) at 24-weeks post-randomization, measured using the patient-reported Edinburgh Postnatal Depression Scale (EPDS). The main secondary outcome is symptom remission (EPDS <10) at 24-weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18 years or older)
2. Pregnant or postpartum and living with their infant 0-6 months old. This includes all individuals who identify as women, as well as those of female sex who do not identify as women (e.g., non-binary, trans) who are the primary parent for their infant. This includes via natural birth, adoption, or surrogacy.
3. EPDS score >10 at eligibility screening.

Exclusion Criteria:

1. Active alcohol or substance use disorder, mania or psychotic disorder (as these conditions are better managed in direct specialty care).
2. Active suicide plan or intent (as emergent hospital-based care is likely required),
3. Plan to move out of Ontario during the study.
4. Unable to complete relevant study procedures and measures online. For the few participants without access to devices/home internet, we will budget for tablets/data plans.
5. Unable to complete study activities in English. Note that Google translate is available for the intervention platform and language lines are available for participants so that they can be served in their language of choice, however we are unable to provide translations of all study assessment and questionnaire materials that participants will need to complete during the study.
6. No primary care clinician (required for collaborative mental health care delivery model).
7. Currently enrolled in a collaborative mental health care model.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 24 weeks post randomization
  The primary objective of this trial is to determine the effect of MOVIN versus a control condition on perinatal depression symptoms. Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30.

SECONDARY OUTCOMES:
Maternal Remission of depression | 24 weeks post randomization
  Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30. A EPDS score of <10 indicates remission.
Maternal Depressive symptoms | 12 weeks post randomization
  Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30.
Maternal Depressive symptoms | 12 and 24 weeks post randomization
  Depressive symptoms will be measured using the Patient Health Questionnaire Scale (PHQ-9), a self-report scale that has been validated for use in pregnancy and postpartum. PHQ-9 scores range from 0 to 27.
Obsessive-Compulsive Inventory-Revised | 12 and 24 weeks post randomization
  OCD symptoms will be measured using the Obsessive-Compulsive Inventory-Revised (OCI-R) Scale, a self-report scale that has been validated for use. OCI-R scores range from 0 to 72.
Maternal Posttraumatic Stress Disorder Checklist | 12 and 24 weeks post randomization
  PTSD symptoms will be measured using the Posttraumatic Stress Disorder Checklist (PCL-5), a self report scale that has been validated to assess for PTSD symptoms. PCL-5 scores range from 0 to 80.
Maternal anxiety symptoms | 12 and 24 weeks post randomization
  Anxiety symptoms will be measured using the General Anxiety Disorder-7 (GAD-7) scale, which is a self-report scale with good discriminate validity in perinatal populations. GAD-7 scores range from 0 to 21, with higher scores indicating more severe symptoms.
Maternal quality of life symptoms | 12 and 24 weeks post randomization
  Quality of life will be measured using the 5 Level-5 Dimension EuroQol 5 (EQ-5D-5L) which is a multi-attribute utility instrument for measuring quality-adjusted life year (QALY), a preference-based utility measure of health-related quality of life as perceived by the patient. It can define 3125 different health states ranging from 11111 (full health) to 55555 (worst health).
Health service use: participant time | 12 and 24 weeks post randomization
  Measured by participant self-report of activities related to attending appointments and obtaining services.
Health service use: participant cost | 12 and 24 weeks post randomization
  Measured by participant self-report of costs related to attending appointments and obtaining services.
Health service use: health system costs | 12 and 24 weeks post randomization
  Calculated from participant self-report of medical costs such as hospitalizations, visits with health professionals and medications.
Maternal child relationship | If postpartum at enrollment: Baseline + 1y postpartum. If pregnant at enrollment: 1y postpartum
  All participants who are postpartum at any time point will complete Parenting Stress Index short form (PSI-SF) to measure parenting stress. This is a 36-item measure consisting of 3 sub-scales: parental distress, dysfunction in the parent-child relations and difficult child. Scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Dyadic relationship | 12 and 24 weeks post randomization
  The Dyadic Adjustment Scale (DAS) is a self-report measure of relationship adjustment with an intimate partner and will be used to measure relationship distress. The first 15 items of the 32-item measure will be used to assess dyadic consensus. Scores range from 0 to 75. Higher scores indicate a higher degree of dyadic consensus.
Child Development | If postpartum at enrollment: Baseline + 1y postpartum. If pregnant at enrollment: 1y postpartum.
  Assessed using the Ages & Stages Questionnaire, Third Edition [ASQ-3 (12 Months)], and the Ages & Stages Questionnaires: Social-Emotional, Second Edition [(ASQ:SE-2 (12 Months)]. A 30-item instrument that screens for child development at 11 months 0 days through 12 months 30 days and 9 months 0 days through 14 months 30 days, respectively. Scores are compared to norms. For the ASQ-3, the minimum value is 0 while the maximum value is 60. For the ASQ:SE-2, The minimum value is 0 while the maximum value is 155. A lower score indicates there may be a concern and further assessment from a professional may be needed, while a higher score indicates no concern and the child's development appears to be on track.

OTHER OUTCOMES:
Clinician perspective survey | 24 weeks post randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No